CLINICAL TRIAL: NCT07396753
Title: The Effects of Transversalis Fascia Plane Block on Opioid Consumption in Patients Undergoing Hand-Assisted Laparoscopic Donor Nephrectomy: A Randomized Controlled Prospective Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Yasemin Sincer, Medical Doctor, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025.030.IRB1.006
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain; Analgesics, Opioid; Pain Management; Anesthesia Regional; Living Donors; Nephrectomy,Kidney Donation
Keywords: Hand-assisted laparoscopic donor nephrectomy; Transversalis fascia plane block; Regional anesthesia; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two separate groups Each participant receives only one intervention Group A: General anesthesia only Group B: General anesthesia + TFPB Outcomes are compared between groups, not within the same patient.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): General anesthesia without regional block
- Group B (Active Comparator): General anesthesia + Ultrasound guided Transversalis Fascia Plane Block (with local anesthetic)
  Interventions: Procedure: Ultrasound-guided transversalis fascia plane block

INTERVENTIONS:
Procedure: Ultrasound-guided transversalis fascia plane block — Ultrasound-guided transversalis fascia plane block performed after induction of general anesthesia using a single-shot injection of 30 mL 0.25% bupivacaine between the posterior surface of the transversus abdominis muscle and the transversalis fascia, targeting T12-L1 thoracolumbar nerve branches (iliohypogastric and ilioinguinal nerves) for postoperative analgesia following hand-assisted laparoscopic donor nephrectomy.
  Arms: Group B

SUMMARY:
This study aims to evaluate whether a regional anesthesia technique called the transversalis fascia plane block (TFPB) can improve pain control after hand-assisted laparoscopic donor nephrectomy (HALDN), a minimally invasive surgery performed in living kidney donors.

Although HALDN is less invasive than open surgery, patients often experience significant pain after the operation, mainly due to the surgical incisions in the lower abdomen and trocar entry sites. Poorly controlled pain can delay recovery and increase the need for opioid pain medications, which may cause side effects such as nausea, vomiting, itching, and sedation.

The transversalis fascia plane block is an ultrasound-guided regional anesthesia technique in which a local anesthetic is injected into a specific tissue plane in the lower abdominal wall. This injection temporarily blocks pain signals from nerves supplying the lower abdomen and groin area. The technique has been shown to reduce pain and opioid use after various lower abdominal surgeries and is considered minimally invasive and safe when performed under ultrasound guidance.

In this study, patients undergoing HALDN will be randomly assigned to one of two groups. One group will receive standard general anesthesia only, while the other group will receive general anesthesia plus a transversalis fascia plane block using a local anesthetic (bupivacaine). All patients will receive the same standard pain treatment after surgery, including paracetamol and patient-controlled morphine.

The main goal of the study is to compare the amount of opioid pain medication used during the first 24 hours after surgery between the two groups. Secondary outcomes include pain scores measured using the Numeric Rating Scale (NRS), the frequency of opioid-related side effects, and patient satisfaction with pain control.

The results of this study may help determine whether adding the transversalis fascia plane block to standard anesthesia can provide better pain relief, reduce opioid consumption, and improve comfort and recovery in living kidney donors.

DETAILED DESCRIPTION:
Study Objective and Hypothesis The primary objective of this prospective, randomized controlled clinical trial is to evaluate the analgesic efficacy of the transversalis fascia plane block (TFPB) in patients undergoing hand-assisted laparoscopic donor nephrectomy (HALDN). The study hypothesizes that the addition of ultrasound-guided TFPB using a local anesthetic will result in lower postoperative opioid consumption and reduced postoperative pain scores, as measured by the Numeric Rating Scale (NRS), during the first 24 hours after surgery.

Background and Rationale HALDN is widely used as a minimally invasive surgical technique for living kidney donation. Despite its minimally invasive nature, postoperative pain remains a significant clinical issue and may negatively affect patient recovery, mobilization, and overall satisfaction. Pain following HALDN is primarily attributed to trocar insertion sites and the lower abdominal incision required for kidney extraction.

Regional anesthesia techniques have increasingly been incorporated into multimodal analgesia strategies to improve postoperative pain control and reduce opioid requirements. However, an optimal regional anesthesia technique for HALDN has not yet been established.

The transversalis fascia plane block is an ultrasound-guided regional anesthesia technique in which local anesthetic is injected between the posterior surface of the transversus abdominis muscle and the transversalis fascia. This approach targets the thoracolumbar nerve branches at the T12-L1 level, including the ilioinguinal and iliohypogastric nerves, which are responsible for sensory innervation of the lower abdominal wall and groin. TFPB has been shown to provide effective analgesia following inguinal hernia repair, lower abdominal surgeries, and urologic procedures.

When performed under ultrasound guidance, TFPB is considered a safe and minimally invasive technique. Potential complications are rare and may include block failure, local anesthetic systemic toxicity, or inadvertent injury to surrounding structures.

Study Design This is a single-center, prospective, randomized controlled trial conducted at Koç University Hospital.

Study Population Eligible participants are adult patients aged 18 to 80 years who have been approved by the transplant committee as living kidney donors and are scheduled for HALDN. Written informed consent will be obtained from all participants prior to enrollment.

Exclusion Criteria Known allergy to any study medications Chronic opioid or opioid receptor agonist use Inability to communicate effectively Presence of chronic organ failure Refusal or inability to provide informed consent Foreign nationality American Society of Anesthesiologists (ASA) physical status classification ≥ III Randomization and Group Allocation

Patients will be randomized using the sealed envelope method into two groups:

Group A (Control Group): General anesthesia only, without any regional anesthesia technique Group B (TFPB Group): General anesthesia plus ultrasound-guided transversalis fascia plane block Anesthesia and Block Technique All patients will undergo standardized general anesthesia. Induction will be achieved with intravenous fentanyl (1-2 µg/kg), propofol (1-2 mg/kg), and rocuronium (0.9-1.2 mg/kg). Maintenance of anesthesia will be provided using oxygen (FiO₂ 35%), desflurane (1 MAC), and continuous intravenous remifentanil infusion (0.02-0.2 µg/kg/min).

In Group B, after induction of general anesthesia and prior to surgical incision, an ultrasound-guided TFPB will be performed using 30 mL of 0.25% bupivacaine. The local anesthetic will be prepared by the anesthesia technician responsible for intraoperative care.

Postoperative Analgesia At the end of surgery, all patients will receive intravenous paracetamol 1 g and morphine 0.05 mg/kg as part of a multimodal analgesia regimen. Neuromuscular blockade will be reversed with sugammadex (200 mg), and patients will be extubated in the operating room before transfer to the post-anesthesia care unit (PACU).

In the PACU, patients with an NRS pain score >4 will receive intravenous fentanyl 50 µg, which may be repeated every 15 minutes, and the total amount will be noted. After stabilization, patients will be transferred to the surgical ward.

Postoperative pain management during the first 24 hours will include routine intravenous paracetamol (1 g three times daily) and patient-controlled analgesia (PCA) with morphine (1 mg bolus, 8-minute lockout, no basal infusion). If pain remains ≥4 on the NRS despite PCA use, intravenous tramadol 50 mg will be administered as rescue analgesia.

Outcome Measures

Primary Outcome:

Total opioid consumption during the first 24 hours after surgery

Secondary Outcomes:

NRS pain scores recorded every 6 hours for 24 hours Incidence of opioid-related side effects (nausea, vomiting, pruritus, allergic reactions) Patient satisfaction with pain management Opioid-related adverse events will be recorded as binary variables (yes/no) every 6 hours.

Statistical Analysis Data will be analyzed using SPSS version 25.0. Continuous variables will be compared using independent t-tests or Mann-Whitney U tests, as appropriate. A p-value <0.05 will be considered statistically significant.

Sample Size Calculation Sample size was determined using power analysis based on institutional data from a previous study evaluating erector spinae plane block in kidney donors, in which 24-hour opioid consumption in the control group was 37.5 ± 18.5 mg. Assuming a 50% reduction in opioid consumption with TFPB, with α = 0.05, β = 0.2, and a completion rate of 90%, a total of 50 patients (25 per group) was calculated to be sufficient. The analysis was performed using G*Power version 3.1.9.7.

ELIGIBILITY:
Inclusion Criteria:

* Approved by the transplant committee for living kidney donation
* Scheduled for hand-assisted laparoscopic donor nephrectomy (HALDN)
* Able to understand study procedures and provide written informed consent

Exclusion Criteria:

* Known allergy to any medications used in the study (e.g., local anesthetics, opioids)
* Chronic opioid use or use of opioid receptor agonists
* Inability to communicate effectively (e.g., cognitive impairment, language barrier)
* Chronic organ failure or major organ dysfunction
* Refusal or inability to provide informed consent
* Foreign nationality (if follow-up or consent is restricted)
* American Society of Anesthesiologists (ASA) physical status ≥ III

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption during the first 24 hours postoperatively | 24 hours after surgery
  Total cumulative opioid consumption (morphine-equivalent dose) within the first 24 hours following hand-assisted laparoscopic donor nephrectomy.

SECONDARY OUTCOMES:
Postoperative pain scores using the Numeric Rating Scale (NRS) | 24 hours postoperatively
  Patient-reported pain intensity on a scale of 0 (no pain) to 10 (worst imaginable pain) at 6, 12, 18, and 24 hours postoperatively.
Incidence of opioid-related adverse effects | 24 hours postoperatively
  Occurrence of nausea, vomiting, pruritus, or allergic reactions, recorded as yes/no at 6, 12, 18, and 24 hours postoperatively.
Rescue analgesic use | Time Frame: 24 hours postoperatively
  The dose of additional analgesics (tramadol 50 mg IV) administered at the surgical ward if NRS for pain is ≥4 despite PCA use.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Gurkan, Prof, Study Director — Koç University Hospital
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include demographic information (age, sex, weight, ASA status), perioperative opioid consumption (morphine-equivalent doses), postoperative pain scores measured by the Numeric Rating Scale (NRS), rescue analgesic use, incidence of opioid-related adverse events (nausea, vomiting, pruritus, allergic reactions), and patient satisfaction with pain management. All shared data will be anonymized to prevent identification of individual participants.
Supporting Information: Study Protocol, ICF
Time Frame: March 2026-March 2031
Access Criteria: Access to the de-identified individual participant data (IPD) and supporting documentation (study protocol, statistical analysis plan, and data dictionary) will be granted to qualified researchers upon reasonable request. Researchers must submit a proposal outlining the objectives of their analysis and obtain approval from the study's principal investigator. Shared data will include de-identified demographic information, perioperative opioid consumption, postoperative NRS pain scores, rescue analgesic use, incidence of opioid-related adverse events, and patient satisfaction scores. Data will be shared in a secure, password-protected format via institutional data-sharing platforms or secure file transfer. All recipients must agree to use the data solely for research purposes and to maintain participant confidentiality.

REFERENCES:
- [Background] Bainton A. Ilioinguinal/iliohypogastric nerve block. Anaesthesia. 1982 Jun;37(6):696-7. doi: 10.1111/j.1365-2044.1982.tb01289.x. No abstract available. PMID 7091630
- [Background] Chen J, Song D, Zheng G, Luo Y. Systematic review and meta-analysis of the effect of nerve block under ultrasound in ilioinguinal/iliohypogastric in children. Transl Pediatr. 2022 Oct;11(10):1604-1614. doi: 10.21037/tp-22-308. PMID 36345442
- [Background] Hamid HKS, Ahmed AY, Alhamo MA, Davis GN. Efficacy and Safety Profile of Rectus Sheath Block in Adult Laparoscopic Surgery: A Meta-analysis. J Surg Res. 2021 May;261:10-17. doi: 10.1016/j.jss.2020.12.003. Epub 2020 Dec 30. PMID 33387729
- [Background] Fleishman A, Khwaja K, Schold JD, Comer CD, Morrissey P, Whiting J, Vella J, Kayler LK, Katz D, Jones J, Kaplan B, Pavlakis M, Mandelbrot DA, Rodrigue JR; KDOC Study Group. Pain expectancy, prevalence, severity, and patterns following donor nephrectomy: Findings from the KDOC Study. Am J Transplant. 2020 Sep;20(9):2522-2529. doi: 10.1111/ajt.15861. Epub 2020 Apr 12. PMID 32185880
- [Background] Zorgdrager M, van Londen M, Westenberg LB, Nieuwenhuijs-Moeke GJ, Lange JFM, de Borst MH, Bakker SJL, Leuvenink HGD, Pol RA. Chronic pain after hand-assisted laparoscopic donor nephrectomy. Br J Surg. 2019 May;106(6):711-719. doi: 10.1002/bjs.11127. Epub 2019 Mar 27. PMID 30919435
- [Background] Gunaydin B, Ucar T, Arpali E, Akyollu B, Akinci S, Karatas C, Oztorun K, Kocak B. Hand-assisted laparoscopic donor nephrectomy: 1864 cases in 15 years of experience. Turk J Med Sci. 2022 Aug;52(4):1322-1328. doi: 10.55730/1300-0144.5438. Epub 2022 Aug 10. PMID 36326419
- [Background] Ozkalayci O, Karakaya MA, Yenigun Y, Cetin S, Darcin K, Akyollu B, Arpali E, Kocak B, Gurkan Y. Effects of erector spinae plane block on opioid consumption in patients undergoing hand-assisted laparoscopic donor nephrectomy: a randomized controlled trial. Minerva Anestesiol. 2024 Mar;90(3):154-161. doi: 10.23736/S0375-9393.23.17706-6. Epub 2024 Feb 2. PMID 38305014